CLINICAL TRIAL: NCT04767672
Title: Randomized, Double-Blinded, Placebo-Controlled Study to Assess the Effects of Short-Chain Fructo-Oligosaccharides on Long-Term Glucose Homeostasis in Untreated Prediabetic Subjects
Brief Title: Study to Assess the Effects of Non Digestible Carbohydrates on Long-Term Glucose Homeostasis in Untreated Prediabetic Subjects
Acronym: FOS_GLUCOSE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tereos (Industry)
Collaborators: BioFortis (Other)
Responsible Party: Principal Investigator, Isabelle Metreau, Coordinating investigator, Tereos
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PEC19095; 2020-A02304-35 (Other: ID-RCB Number)
Record Dates: First submitted 2021-02-19; First posted 2021-02-23 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Pre Diabetes; Prediabetic State; Dysglycemia; PreDiabetes
MeSH Terms: conditions — Glucose Intolerance; Prediabetic State

STUDY DESIGN:
Intervention Model Description: multicentre randomized, parallel arms, double-blind, placebo-controlled clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test product (Experimental): Food ingredient containing non digestible carbohydrates, in shape of powder
  Interventions: Dietary Supplement: Non digestible carbohydrates
- Placebo (Placebo Comparator): Food ingredient containing containing 95% of maltodextrin
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Non digestible carbohydrates — the subjects will consume 2 bags of 10 grams per day of the product: 1 bag in the morning and 1 bag at lunch or in the evening, at the beginning of the meal, diluted in a large glass of beverage, during 12 weeks.
  Arms: Test product
Dietary Supplement: Placebo — the subjects will consume 2 bags of 10 grams per day of the product: 1 bag in the morning and 1 bag at lunch or in the evening, at the beginning of the meal, diluted in a large glass of beverage, during 12 weeks.
  Arms: Placebo

SUMMARY:
This clinical study aims to prove that the efficacy of non digestible carbohydrates supplementation (daily dose of 20 grams consumed twice a day for 12 weeks) on the regulation of glucose homeostasis is superior than placebo in prediabetic subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years (limits included);
* BMI between 23 and 34.9 kg/m² (limits included);
* Dysglycemic or prediabetic subjects with no antidiabetic medication (medical or lifestyle (hygiene-dietetic measures or specific regimen treatment);
* Consuming 10 to 20 g quantity of fiber per day (based on the 3-days food diary fulfilled by the subject between V1 and V2 visits);
* Smoking maximum 10 cigarettes per week or equivalent and agreeing to keep this habit unchanged throughout the study;
* Able and willing to participate to the study by complying with the protocol procedures as evidenced by his dated and signed informed consent form;
* Affiliated with a social security scheme;
* Agree to be registered on the volunteers in biomedical research file;
* Fasting venous glycemia ≥ 1 g/L and ≤ 1.25 g/L at V1 visit.

Exclusion Criteria:

* Metabolic disorder such as diabetes, uncontrolled thyroidal trouble or other metabolic disorder;
* Severe chronic disease or Intestinal Bowel Syndrome (IBS) or gastrointestinal disorders found to be inconsistent with the conduct of the study by the investigator;
* History of retinopathy, microalbuminuria, ischemic cardiovascular event in the 6 months before the study;
* Known or a suspected food allergy or intolerance orhypersensitivity to any food ingredient;
* Known or suspected food allergy or intolerance or hypersensitivity to any of the study products' ingredient;
* Pregnant or lactating women or intending to become pregnant within 4 months ahead;
* Women starting hormone replacement therapy or oral contraception (treatment must be stable for at least 3 months);
* History of bariatric surgery;
* History of any surgery in the 3 months before V1 visit or having scheduled any surgery within 4 months ahead;
* Under dietary supplement which could significantly affect parameter(s) followed during the study according to the investigator or stopped in a too short period before the V1 visit (< 3 months);
* Under treatment which could significantly affect parameter(s) followed during the study according to the investigator or stopped less than 3 months before the V1 visit;
* Under antibiotic treatment in the 3 to 6 months before V1 visit, depending on the antibiotic consumed and according to the investigator;
* Significant change in food habits or in physical activity in the 3 months before V1 visit or not agreeing to keep them unchanged throughout the study;
* Current or planned in the next 4 months specific diet (hyper or hypocaloric, vegan, vegetarian…) or stopped less than 3 months before the study;
* Personal history of anorexia nervosa, bulimia or significant eatingdisorders according to the investigator;
* Consuming more than 3 standard drinks of alcoholic beverage daily for men or 2 daily for women or not agreeing to keep his alcohol consumption habits unchanged throughout the study;
* Taking part in another clinical trial or being in the exclusion period of a previous clinical trial;
* Having received, during the last 12 months, indemnities for clinical trial higher or equal to 4500 Euros;
* Under legal protection (guardianship, wardship) or deprived from his rights following administrative or judicial decision;
* Psychological or linguistic incapability to sign the informed consent;
* Impossible to contact in case of emergency.
* Fasting blood triglycerides > 3,5 g/L;
* Fasting blood of total cholesterol > 4,5 g/L or HDLc < 0,1 g/L with an abnormality judged as clinically significant according to the investigator;
* Blood ASAT, ALAT or GGT > 3 times ULN (laboratory Upper Limit of Normal);
* Blood urea > 12 mmol/L or creatinine > 125 μmol/L;
* Complete Blood Count (CBC) with hemoglobin < 11 g/L or leucocytes < 3000/mm3 or leucocytes > 16000/mm3.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Glycated hemoglobin | V2 (randomization) and V5 (12 weeks of intervention)
  Change from baseline of Hba1c level (%)

SECONDARY OUTCOMES:
Glycated hemoglobin | V2 (randomization), V3 (4 weeks of intervention), V4 (8 weeks of intervention) and V5 (12 weeks of intervention)
  Absolute variations of Hba1c level (%)
Fasting glycemia | V2 (randomization), V3 (4 weeks of intervention), V4 (8 weeks of intervention) and V5 (12 weeks of intervention)
  Change from baseline of fasting glycemia (g/L)
Fasting insulinemia | V2 (randomization), V3 (4 weeks of intervention), V4 (8 weeks of intervention) and V5 (12 weeks of intervention)
  Change from baseline of fasting insulinemia (mU/L)
Fructosamine | V2 (randomization), V3 (4 weeks of intervention), V4 (8 weeks of intervention) and V5 (12 weeks of intervention)
  Change from baseline of fructosamine (μmol/L)
Insulin indexes | V2 (randomization), V3 (4 weeks of intervention), V4 (8 weeks of intervention) and V5 (12 weeks of intervention)
  Change from baseline of HOMA-IR (Homeostasis Model Assessment of Insulin) and QUICKI (Quantitative Insulin sensitivity Check Index) indices
Insulin sensitivity index | V2 (randomization) and V5 (12 weeks of intervention)
  Change from baseline of insulin sensitivity index (ISI)
Glycemia level | V2 (randomization) and V5 (12 weeks of intervention)
  Change from baseline of glycemia level (g/L)
Incremental Area Under the Curve (iAUC) of glycemia | V2 (randomization) and V5 (12 weeks of intervention)
  Change from baseline of iAUC of glycemia (g/L)
Insulinemia | V2 (randomization) and V5 (12 weeks of intervention)
  Change from baseline of insulinemia levels (mU/L)
Incremental Area Under the Curve (iAUC) of insulinemia | V2 (randomization) and V5 (12 weeks of intervention)
  Change from baseline of iAUC of insulinemia (mU/L)
Glucacon-like Peptide 1 (GLP-1) | V2 (randomization) and V5 (12 weeks of intervention)
  Change from baseline of GLP-1 levels (pmol/L)
Bone mineral composition | V2 (randomization) and V5 (12 weeks of intervention)
  Change from baseline of bone mineral composition (kg)
Total lean mass | V2 (randomization) and V5 (12 weeks of intervention)
  Change from baseline of total lean mass (g and %)
Total fat mass | V2 (randomization) and V5 (12 weeks of intervention)
  Change from baseline of total fat mass (g and %)
Bone Mineral Density | V2 (randomization) and V5 (12 weeks of intervention)
  Change from baseline of bone mineral density (g/cm2)
Total Body Mass | V2 (randomization) and V5 (12 weeks of intervention)
  Change from baseline of total body mass (kg)
Weight | V2 (randomization), V3 (4 weeks of intervention), V4 (8 weeks of intervention) and V5 (12 weeks of intervention)
  Change from baseline of weight (in kg)
Body Mass Index (BMI) | V2 (randomization), V3 (4 weeks of intervention), V4 (8 weeks of intervention) and V5 (12 weeks of intervention)
  Change from baseline of BMI (in kg/m2)
Waist and Hip measurement | V2 (randomization), V3 (4 weeks of intervention), V4 (8 weeks of intervention) and V5 (12 weeks of intervention)
  Change from baseline of waist and hip Circumference (in cm)
Anthropometric ratios | V2 (randomization), V3 (4 weeks of intervention), V4 (8 weeks of intervention) and V5 (12 weeks of intervention)
  Change from baseline of Waist to Hip ratio and Waist to Height ratio
Satiety and Appetite sensation | V2 (randomization) and V5 (12 weeks of intervention)
  Change on satiety and appetite sensation using 100-mm VAS to complete 15 min before the meal, 30 min, 60 min, 120 min, 180 min and 240 min after the meal at which study product was consumed
Total energy intake | V2 (randomization), V3 (4 weeks of intervention), V4 (8 weeks of intervention) and V5 (12 weeks of intervention)
  Change from baseline of total energy intake - TEI (kcal/day)
Energy intake | V2 (randomization), V3 (4 weeks of intervention), V4 (8 weeks of intervention) and V5 (12 weeks of intervention)
  Change from baseline of percentage of energy intake from fat, carbohydrates and protein (g and %TEI)
Fiber intake | V2 (randomization), V3 (4 weeks of intervention), V4 (8 weeks of intervention) and V5 (12 weeks of intervention)
  Change from baseline of percentage of percentage of fiber (g)
Alcohol intake | V2 (randomization), V3 (4 weeks of intervention), V4 (8 weeks of intervention) and V5 (12 weeks of intervention)
  Change from baseline of percentage of percentage of alcohol intake (absolute quantities, g/day)
Biomarker of inflammation | V2 (randomization), V3 (4 weeks of intervention), V4 (8 weeks of intervention) and V5 (12 weeks of intervention)
  Change from baseline of high-sensitivity C-reactive Protein (CRPhs) (mg/L)
Intestinal microbiota composition | V2 (randomization) and V5 (12 weeks of intervention)
  Change from baseline microbiota composition for alpha-diversity indices (Shannon and Chao indices) and abundances at the phylum, family and genus level assessed by 16S metabarcoding (in a subgroup of 30 subjects only)
Fecal Short-Chain Fatty Acids (SCFA) | V2 (randomization) and V5 (12 weeks of intervention)
  Change from baseline of fermentative activity of the intestinal microbiota assessed by measuring short-chain fatty acids concentrations in stool (in the same subgroup of 30 subjects only)

OTHER OUTCOMES:
Incidence of adverse events (AEs) | V1 (Inclusion), V2 (randomization), V3 (4 weeks of intervention), V4 (8 weeks of intervention) and V5 (12 weeks of intervention)
  Number of adverse events (including gastro-intestinal symptoms) by subject that appeared during the entire duration of the study
Heart Rate (HR) | V2 (randomization), V3 (4 weeks of intervention), V4 (8 weeks of intervention) and V5 (12 weeks of intervention)
  Change from baseline of HR (bpm)
Blood pressure | V2 (randomization), V3 (4 weeks of intervention), V4 (8 weeks of intervention) and V5 (12 weeks of intervention)
  Change from baseline of Systolic Blood Pressure and Diastolic Blood Pressure (mmHg)

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - IPL, Lille
  - Biofortis Center Paris, Paris
  - UIC BIOFORTIS Saint-Herblain, Saint-Herblain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Le Bourgot C, Capronnier O, Graf S, Carton T. Targeting gut microbiota with short-chain fructo-oligosaccharides prebiotic fibers to support metabolic health in overweight prediabetic adults: a randomized, double-blinded, placebo-controlled study. Front Nutr. 2025 Dec 17;12:1718169. doi: 10.3389/fnut.2025.1718169. eCollection 2025. PMID 41479657